CLINICAL TRIAL: NCT01187485
Title: A Randomized Phase I Study of Testosterone Replacement in Patients With Low Risk Hormone Refractory Prostate Cancer
Brief Title: A Randomized Study of Testosterone Replacement in Patients With Low Risk Hormone Refractory Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13183B
Record Dates: First submitted 2010-08-20; First posted 2010-08-24 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Prostate Cancer
Keywords: Androderm®; Testosterone; refractory; prostate; cancer; Patients with "hormone refractory" prostate cancer will be treated with a daily testosterone patch Androderm® applied every 24 hours to the skin
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Androderm® 2.5mg (Experimental): Study subjects will be randomized to one of the study arms: 2.5 mg of Androderm®.
  Interventions: Drug: Androderm® 2.5mg
- Androderm® 5.0 mg (Experimental): Study subjects will be randomized to one of the study arms: 5.0 mg of Androderm®.
  Interventions: Drug: Androderm® 5.0mg
- Androderm® 7.5mg (Experimental): Study subjects will be randomized to one of the study arms: 7.5 mg of Androderm®.
  Interventions: Drug: Androderm® 7.5mg

INTERVENTIONS:
Drug: Androderm® 2.5mg — Subjects will be asked to replace the study drug patch every 24 hours at night following the written and verbal instructions you will receive. The study drug patch should be placed over a small amount of a steroid cream on the skin to reduce irritation.
  Arms: Androderm® 2.5mg
Drug: Androderm® 5.0mg — Subjects will be asked to replace the study drug patch every 24 hours at night following the written and verbal instructions you will receive. The study drug patch should be placed over a small amount of a steroid cream on the skin to reduce irritation.
  Arms: Androderm® 5.0 mg
Drug: Androderm® 7.5mg — Subjects will be asked to replace the study drug patch every 24 hours at night following the written and verbal instructions you will receive. The study drug patch should be placed over a small amount of a steroid cream on the skin to reduce irritation.
  Arms: Androderm® 7.5mg

SUMMARY:
The purpose of this study is to see how safe Androderm® (the study drug) is at three different doses in subjects with early hormone refractory prostate cancer. In addition, information about hormonal levels and the effects of testosterone on quality of life including sexual functioning and muscle strength will be collected.

DETAILED DESCRIPTION:
Most hormone-refractory disease is currently defined by rising PSA following androgen ablation and an antiandrogen. These patients are typically asymptomatic and have minimal or no radiologically evident disease by standard bone and CT scans. Therapeutic options are limited, with 3rd line hormonal treatments generally providing only brief durations of benefit in a small minority of patients. Chemotherapy is effective, but the role of this somewhat toxic approach in the asymptomatic patient is debatable. In addition, patients suffer from the long-term side effects of androgen ablation such as muscle wasting, decreased strength, decreased sexual functioning, and impaired cognition. If the hypothesis that androgen replacement can inhibit cancer growth in androgen insensitive patients is correct, such treatment would not only delay disease progression but could also improve quality of life. If the hypothesis is incorrect and androgens actually stimulate growth, the consequences are unlikely to be catastrophic since the selected population has only a minimal disease burden.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a histologically documented diagnosis of prostate adenocarcinoma (PCa) not amenable to curative treatment with surgery or radiation treatment.
* Patient was surgically or pharmacologically castrated at least 6 months prior to randomization. Castration must be verified by a screening testosterone value of <30 ng/dL. Any patient pharmacologically castrated must be maintained on androgen suppression therapy for the duration of the study.
* Patient must have had a previous trial of anti-androgen therapy.
* Patients must have a documented anti-androgen withdrawal period prior to randomization: flutamide requires a minimum 4 weeks withdrawal, and nilutamide and bicalutamide require a minimum 6 weeks withdrawal.
* Patient must meet one of the following PSA criteria:
* A 50% rise in PSA values within a minimum rise to at least 3.0 ng/mL, within 6 months prior to randomization, OR
* A rising PSA defined as two sequential increases in PSA values. The following data are required: an initial value (#1) followed by a PSA value demonstrating an increase (#2). The increase must be confirmed by another rise in PSA (#3) (3>2>1). There must be at least 2 weeks between each qualifying PSA value and the absolute PSA value at enrollment must be at least 3.0 ng/ml.
* At the time of screening the patient must have no evidence of visceral organ-confined metastatic disease OR the presence of minimal bone metastases only without evidence of visceral organ-confined metastatic disease.
* The absence of visceral organ-confined metastatic disease is defined as:

  * No organ-confined soft tissue metastases (e.g. lung, liver, etc.) as verified by chest/abdomen/pelvic CT scan.
* The presence of pathologically enlarged lymph nodes will not exclude subjects from the study and will not be included in the definition of visceral organ-confined metastatic disease.
* The presence of minimal bone metastases is defined as <1.4% by Bone Scan Index criteria (see section 9).
* ECOG performance status <2 (Karnofsky >70%, see Appendix A).
* Age >18 years. Because no dosing or adverse event data are currently available on the use of Androderm® in the context of androgen ablation in patients <18 years of age, children are excluded from this study but will be eligible for future pediatric phase 1 single-agent trials.
* Patients must have normal hepatic and renal function as defined below:
* total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) <1.5 X institutional upper limit of normal
* Patient has had no other active malignancies with the exception of non-melanoma skin cancer.
* Patient must possess the ability to understand and be willing to sign a written informed consent document.

Exclusion Criteria:

* Patients with a history of any previous cytotoxic therapy or radionuclide therapy (such as rhenium, strontium, or samarium).
* Patients may not be receiving any other investigational agents.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with evidence of visceral organ-confined metastases other than minimal bone metastases (as defined by <1.4% Bone Scan Index, see section 9) and/or pathologically enlarged lymph nodes will be excluded.
* Patients with local recurrences who are candidates for local salvage therapy (e.g. surgery, radiation, brachytherapy, cryotherapy) will be excluded.
* Patients with significant pulmonary disease who have received chronic or pulse steroid therapy within the last 3 months prior to randomization will be excluded. Steroid therapy for non-pulmonary, non-oncologic conditions are allowed if the patient has been on a chronic, steady-dose regimen for a minimum of 2 months prior to randomization.
* Patients with known skin allergies to polyester, alcohol, aluminum, or silicone.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2004-06; Primary Completion 2008-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Primary Study Objective is to determine the safety of Androderm® 2.5 mg, 5.0 mg, and 7.5 mg in patients with early hormone refractory prostate cancer. | 1-4 years
  To determine the safety of Androderm® 2.5 mg, 5.0 mg, and 7.5 mg in patients with early hormone refractory prostate cancer.

SECONDARY OUTCOMES:
Secondary Study Objectives are to determine the effects of Androderm® 2.5 mg, 5.0 mg, and 7.5 mg on total and free testosterone levels and PSA as well as on QOL, sexual functioning, and muscle strength. | 3-5 years
  To determine the effects of Androderm® 2.5 mg, 5.0 mg, and 7.5 mg on total and free testosterone levels and PSA. To determine the effects of Androderm® 2.5 mg, 5.0 mg, and 7.5 mg on QOL, sexual functioning, and muscle strength.

CONTACTS AND LOCATIONS:
Overall Officials: Walter M Stadler, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States